CLINICAL TRIAL: NCT00583375
Title: A Prospective, Randomized, Controlled, Multi-Center, Pivotal Human Clinical Trial to Evaluate the Safety and Effectiveness of Augment® Bone Graft Compared to Autologous Bone Graft as a Bone Regeneration Device in Foot and Ankle Fusions
Brief Title: Augment® Bone Graft (Formerly GEM OS™1 Bone Graft) Compared to Autologous Bone Graft in Foot and Ankle Fusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioMimetic Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMTI-2006-01
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Foot Fusion
Keywords: arthritis; ankle pain; foot pain; hindfoot fracture; ankle fracture
MeSH Terms: conditions — Arthritis; Ankle Fractures | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Standard Rigid Fixation plus autograft
  Standard of Care: Autologous Bone Graft
  Interventions: Procedure: Standard of Care
- Group 2 (Experimental): Standard Rigid Fixation plus Augment® Bone Graft
  Interventions: Device: Augment® Bone Graft

INTERVENTIONS:
Device: Augment® Bone Graft — Augment® Bone Graft
  Arms: Group 2
Procedure: Standard of Care — Autologous Bone Graft
  Arms: Group 1

SUMMARY:
STUDY OBJECTIVES: Demonstrate equivalent clinical and radiologic outcomes to the "gold standard" (ABG) in a representative clinical model (hindfoot and ankle fusions)

STUDY HYPOTHESIS: Augment® Bone Graft is an equivalent bone grafting substitute to autologous bone graft in applications as shown by non-inferiority analysis

STUDY RATIONALE: Evaluate a fully synthetic growth-factor enhanced bone graft substitute to facilitate fusion in conditions or injuries requiring bone graft in a representative clinical fusion model and thus the opportunity to provide equivalent union rates as ABG without necessitating an additional invasive procedure to harvest the graft

REGULATORY PHASE: Investigational Device Exemption (IDE) for Premarket Approval (PMA) Application as a bone regeneration system, pivotal phase

ELIGIBILITY:
Inclusion Criteria:

1) Bone defect in the hindfoot or ankle requiring fusion using open surgical technique with supplemental bone graft/substitute, requiring one of the following procedures:

* Ankle joint fusion
* Subtalar fusion
* Calcaneocuboid fusion
* Talonavicular fusion
* Triple arthrodesis (subtalar, talonavicular and calcaneocuboid joints)
* Double fusions (talonavicular and calcaneocuboid joints)

Exclusion Criteria:

1. Previous fusion surgery of the proposed fusion site.
2. The patient uses chronic medications known to affect the skeleton (e.g. glucocorticoid usage > 10mg/day).
3. Pregnant or a female intending to become pregnant during this study period.
4. Morbidly obese (BMI > 45 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2007-04; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher DiGiovanni, M.D., Principal Investigator — Rhode Island Hospital
Locations (37):
- United States (31):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - California Pacific Orthopaedics & Sports Medicine, San Francisco, California
  - Santa Cruz Orthopaedic Institute, Santa Cruz, California
  - Hartford Hospital Orthopaedic Center, Hartford, Connecticut
  - The Center for Bone & Joint Surgery, Royal Palm Beach, Florida
  - Southern Orthopaedic Center, Savannah, Georgia
  - Illinois Bone and Joint Institute, Ltd., Glenview, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Advanced Orthopaedic Associates, Wichita, Kansas
  - Union Memorial Hospital, Baltimore, Maryland
  - Mid Michigan Orthopaedic Institute, East Lansing, Michigan
  - Orthopaedic Associates of Grand Rapids, Grand Rapids, Michigan
  - Henry Ford Hospital - West Bloomfield, West Bloomfield, Michigan
  - Desert Orthopaedic Center, Las Vegas, Nevada
  - UMDNJ, Newark, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Ortho Carolina Research Institute, Charlotte, North Carolina
  - Duke Health Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Orthopedic Foot & Ankle Center, Columbus, Ohio
  - Orthopaedic & Neurosurgical Care & Research, Bend, Oregon
  - The Rothman Institute, Philadelphia, Pennsylvania
  - University Orthopaedics, Inc, Providence, Rhode Island
  - Campbell Clinic, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Bone and Joint Clinic of Houston, Houston, Texas
  - The Orthopaedic Foot and Ankle Center, Arlington, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (6):
  - Peter Lougheed Centre, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 subjects excluded post-operatively
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 142 | 272
Completed | 142 | 272
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of 414 patients, 272 randomized to Augment® Bone Graft and 142 randomized to autograft. The mITT population, submitted as the primary effectiveness analysis for the radiographic evaluation of bridging bone, consisted of 397 patients (414 patients in the Safety group minus 17 subjects excluded post-operatively).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 142 | 272 | 414
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (13.4) | 55.9 (14.5) | 56.47 (14.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 143 | 204
  Male | 81 | 129 | 210
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 19 | 25
  White | 131 | 247 | 378
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 32 | 67 | 99
  United States | 110 | 205 | 315

OUTCOME MEASURES:

1. Primary Outcome: Subjects Fused at 24 Weeks (as Determined by CT Assessment)
Description: An independent radiologist examined CT images for all patients' joints and determined whether or not the joint had at least 50% osseous bridging. If a patient demonstrated all joints having at least 50% osseous bridging, this patient was classified as fused.
Time Frame: 24 weeks
Population: The mITT population consisted of 397 patients (414 patients in the Safety group minus 17 subjects excluded post-operatively).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 137 | 260
Participants | 85 | 159

2. Secondary Outcome: Pain on Weight Bearing
Description: Subjects were asked to stand and report pain on a 100 mm Visual Analog Scale (with 0 being no pain and 100 being worst pain imaginable).
  1. Clinically significant improvement: ≥20mm decrease from baseline
  2. Detectable improvement: 10-20mm decrease from baseline
  3. Maintained: <10mm decrease from baseline and <10mm increase from baseline
  4. Deteriorated: >10mm increase from baseline
Time Frame: 24 and 52 Weeks
Population: Analysis conducted on patients at 24 and 52 weeks time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 118 | 219
Participants
  Clinically Significant Improvement at 24 weeks: number analyzed (Participants) | 117 | 219
  Clinically Significant Improvement at 24 weeks | 87 | 167
  Detectable Improvement at 24 weeks: number analyzed (Participants) | 117 | 219
  Detectable Improvement at 24 weeks | 12 | 14
  Maintained at 24 weeks: number analyzed (Participants) | 117 | 219
  Maintained at 24 weeks | 12 | 25
  Deteriorated at 24 weeks: number analyzed (Participants) | 117 | 219
  Deteriorated at 24 weeks | 6 | 13
  Clinically Significant Improvement at 52 weeks: number analyzed (Participants) | 118 | 215
  Clinically Significant Improvement at 52 weeks | 95 | 170
  Detectable Improvement at 52 weeks: number analyzed (Participants) | 118 | 215
  Detectable Improvement at 52 weeks | 8 | 20
  Maintained at 52 weeks: number analyzed (Participants) | 118 | 215
  Maintained at 52 weeks | 11 | 19
  Deteriorated at 52 weeks: number analyzed (Participants) | 118 | 215
  Deteriorated at 52 weeks | 4 | 6

3. Secondary Outcome: Pain at Fusion Site
Description: Subjects were asked to report current pain level at the fusion site on a 100 mm Visual Analog Scale (with 0 being no pain and 100 being worst pain imaginable).
  1. Clinically significant improvement: ≥20mm decrease from baseline
  2. Detectable improvement: 10-20mm decrease from baseline
  3. Maintained: <10mm decrease from baseline and <10mm increase from baseline
  4. Deteriorated: >10mm increase from baseline
Time Frame: 24 and 52 weeks
Population: Analysis conducted on patients at 24 and 52 weeks time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 120 | 223
Participants
  Clinically Significant Improvement at 24 weeks | 71 | 144
  Detectable Improvement at 24 weeks | 15 | 20
  Maintained at 24 weeks | 21 | 39
  Deteriorated at 24 weeks | 10 | 20
  Clinically Significant Improvement at 52 weeks: number analyzed (Participants) | 120 | 218
  Clinically Significant Improvement at 52 weeks | 81 | 139
  Detectable Improvement at 52 weeks: number analyzed (Participants) | 120 | 218
  Detectable Improvement at 52 weeks | 11 | 27
  Maintained at 52 weeks: number analyzed (Participants) | 120 | 218
  Maintained at 52 weeks | 19 | 44
  Deteriorated at 52 weeks: number analyzed (Participants) | 120 | 218
  Deteriorated at 52 weeks | 9 | 8

4. Secondary Outcome: Foot Function Index (FFI)
Description: The Foot Function Index (FFI) measures the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales. To obtain a sub-scale score, the item scores for a sub-scale are totaled and then divided by the maximum total possible for all of the sub-scale items which the subject indicated were applicable. Any item marked as not applicable is excluded from the total possible. Sub-scales are an average of the completed ratings within that sub-scale. The total foot function score is an average of the three sub-scale scores. Lower scores are indicative of better outcomes whereas higher scores indicate greater impairment.
  1. Clinically significant improvement: ≥10 point decrease from baseline
  2. Improved: 5-10 point decrease from baseline
  3. Maintained: <5 point decrease from baseline and <5 point increase from baseline
  4. Deteriorated: >5 point increase from baseline
Time Frame: 24 and 52 weeks
Population: Analysis conducted on patients at 24 and 52 weeks time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 133 | 249
Participants
  Clinically Significant Improvement at 24 weeks | 106 | 190
  Improved at 24 weeks | 4 | 19
  Maintained at 24 weeks | 14 | 16
  Deteriorated at 24 weeks | 9 | 24
  Clinically Significant Improvement at 52 weeks: number analyzed (Participants) | 132 | 241
  Clinically Significant Improvement at 52 weeks | 114 | 209
  Improved at 52 weeks: number analyzed (Participants) | 132 | 241
  Improved at 52 weeks | 1 | 8
  Maintained at 52 weeks: number analyzed (Participants) | 132 | 241
  Maintained at 52 weeks | 12 | 12
  Deteriorated at 52 weeks: number analyzed (Participants) | 132 | 241
  Deteriorated at 52 weeks | 5 | 12

5. Secondary Outcome: AOFAS Hindfoot and Ankle Score
Description: Subjects were asked to report pain, functionality and ability levels while the physician performed assessments based on alignment, abnormality, motion, and stability. The total score ranges from a low of zero to a high of 100, with subscales measuring pain (40 points), function (50 points), and alignment (10 points), with higher scores showing better outcomes.
  1. Clinically significant improvement: ≥20 point increase from baseline
  2. Improved: 10-20 point increase from baseline
  3. Maintained: <10 point increase from baseline and <10 point decrease from baseline
  4. Deteriorated: >10 point decrease from baseline
Time Frame: 24 and 52 weeks
Population: Analysis conducted on patients at 24 and 52 weeks time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 133 | 249
Participants
  Clinically Significant Improvement at 24 weeks: number analyzed (Participants) | 133 | 248
  Clinically Significant Improvement at 24 weeks | 94 | 180
  Improved at 24 weeks: number analyzed (Participants) | 133 | 248
  Improved at 24 weeks | 19 | 27
  Maintained at 24 weeks: number analyzed (Participants) | 133 | 248
  Maintained at 24 weeks | 14 | 35
  Deteriorated at 24 weeks: number analyzed (Participants) | 133 | 248
  Deteriorated at 24 weeks | 6 | 8
  Clinically Significant Improvement at 52 weeks: number analyzed (Participants) | 132 | 241
  Clinically Significant Improvement at 52 weeks | 106 | 195
  Improved at 52 weeks: number analyzed (Participants) | 132 | 241
  Improved at 52 weeks | 10 | 22
  Maintained at 52 weeks: number analyzed (Participants) | 132 | 249
  Maintained at 52 weeks | 11 | 19
  Deteriorated at 52 weeks: number analyzed (Participants) | 132 | 249
  Deteriorated at 52 weeks | 5 | 5

6. Secondary Outcome: SF-12 Physical Component Score
Description: The SF-12 Physical Component Score is a validated quality of life metric with a minimum of zero and a maximum of 100, with higher scores denoting higher quality of life.
  1. Maintenance or improvement: ≥0 point increase from baseline
  2. Slight Decline: 0-10 point decrease from baseline
  3. Deteriorated: >10 point decrease from baseline
Time Frame: 24 and 52 weeks
Population: Analysis conducted on patients at 24 and 52 weeks time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 133 | 249
Participants
  Maintenance or Improvement at 24 weeks | 106 | 203
  Slight Decline at 24 weeks | 22 | 38
  Deteriorated at 24 weeks | 5 | 8
  Maintenance or Improvement at 52 weeks: number analyzed (Participants) | 132 | 241
  Maintenance or Improvement at 52 weeks | 117 | 206
  Slight Decline at 52 weeks: number analyzed (Participants) | 132 | 241
  Slight Decline at 52 weeks | 14 | 33
  Deteriorated at 52 weeks: number analyzed (Participants) | 132 | 241
  Deteriorated at 52 weeks | 1 | 2

ADVERSE EVENTS:
Time Frame: Patients were assessed through study completion scheduled at 52 weeks following surgery.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/142 | 1/272
Serious Adverse Events (participants affected / at risk) | 21/142 | 28/272
Other Adverse Events (participants affected / at risk) | 43/142 | 100/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=142) | Group 2 (N=272)
Acute myocardial infarction (Cardiac disorders) | 3 (4) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Congenital foot malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (3)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 2 (2)
Not -cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Device related infection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical device complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound infection staphylococcal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Prothrombin level abnormal (Investigations) | 0 (0) | 1 (1)
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Osteotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic steonsis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 4 (4)
Pulmonary embolism (Vascular disorders) | 1 (1) | 3 (3)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=142) | Group 2 (N=272)
Medical device pain (Injury, poisoning and procedural complications) | 7 (7) | 14 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (17) | 38 (46)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 (24) | 48 (56)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes